CLINICAL TRIAL: NCT02880319
Title: Phase II Protocol Evaluating Stereotactic Body Radiation Therapy for Oligometastatic Disease of the Bone
Brief Title: Evaluating Stereotactic Body Radiation Therapy for Oligometastatic Disease of the Bone
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Tracy Balboni, MD, MPH, Tracy Balboni, MD, MPH, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-207
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Results first posted 2023-08-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Bone Cancer
Keywords: Bone Cancer
MeSH Terms: conditions — Bone Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oligometastatic Disease (Experimental): Stereotactic Body Radiation Therapy (SBRT)to up to 3 sites of disease occurring in the bone or spine
  * Treatments will be delivered on a dedicated stereotactic linear accelerator that includes onboard conebeamCT imaging and orthogonal 2D/3D matching with robotic couch top.
  * Dosage will be determined by physician
  Interventions: Drug: Stereotactic Body Radiation Therapy (SBRT); Device: Stereotactic Linear Accelerator
- Re-irradiation to Metastatic Disease (Experimental): Stereotactic Body Radiation Therapy (SBRT) to site(s) of disease occurring in the bone or spine
  * Treatments will be delivered on a dedicated stereotactic linear accelerator that includes onboard conebeamCT imaging and orthogonal 2D/3D matching with robotic couch top.
  * Dosage will be determined by physician
  Interventions: Drug: Stereotactic Body Radiation Therapy (SBRT); Device: Stereotactic Linear Accelerator

INTERVENTIONS:
Drug: Stereotactic Body Radiation Therapy (SBRT)
Device: Stereotactic Linear Accelerator

SUMMARY:
This research study is studying a form of radiation therapy called stereotactic body radiation therapy or SBRT as a possible treatment for Cancer that has spread to the spine or other bone

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating metastases of the bone. "Investigational" means that the intervention is being studied.

SBRT is an advanced technique that allows for more precise delivery of radiation than with standard radiation therapy. In comparison to standard radiation therapy, it allows us to give higher doses of radiation to a tumor while limiting the radiation dose going to the surrounding normal tissues. This technology has been made possible by advances in imaging and treatment capabilities on the radiation treatment machines. SBRT works just as standard radiation therapy works by damaging cancer cells.

SBRT has been used to deliver radiation to people with cancer in the lung and those with metastases in the spine or liver. Studies of those groups have shown low rates of side effects with good rates of killing the cancer in that area and preventing it from coming back. In the current research study, the investigators are looking to further evaluate how well this type of radiation controls disease in bone and whether the toxicity (side effects) of SBRT differs from that of standard treatment. The investigators hypothesis is that toxicity might be less, as less normal tissue receives radiation with SBRT than with standard treatment. It is important to note that SBRT, just like standard radiation therapy for the participant disease, is being used to attempt to stop the growth of cancer cells in a bone metastasis and relieve or prevent any symptoms (ex. pain) associated with bone metastases. The goal of the SBRT is not to cure the participant cancer. The primary goal of the study is to see how well SBRT controls the disease in the bone, and the investigators also want to analyze its ability to control disease symptoms without added toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Both cohorts:

  --≥18 years of age
  * ECOG performance status ≤2
  * Pathologically proven metastatic solid tumor (non-hematologic malignancy) of the bone (spine or non-spine bone)
  * Bony metastatic lesions must be ≤6 cm in maximum dimension and evaluable on either a CT or MRI scan; metastatic lesions in the spine must involve ≤3 contiguous vertebral bodies
  * No other active malignancy within the past 2 years, except for non-melanoma skin cancers or carcinoma in situ of the cervix
  * Ability to understand and the willingness to sign a written informed consent document
  * Surgery to the lesion in question is allowed if size criteria outlined above are met
  * Not currently pregnant or breast feeding
* Cohort 1: Oligometastatic state

  * Oligometastatic state is defined by ≤ 3 active sites of disease, including the primary site
  * Agreement of both the Chow et al.15 and TEACHH16 models, indicating a median life expectancy of >3 months
  * Among patients with multiple sites of metastatic disease, the other sites that will not be treated on this protocol have either been previously treated or are planned for local treatment
* Cohort 2: Re-irradiation

  * Previous radiation in the current area of disease requiring radiation
  * Life expectancy of >3 months as defined by agreement of both the Chow et al.15 and TEACHH16 models

Exclusion Criteria:

* SBRT target size >6 cm in maximum diameter (or >100 cc in volume)
* Hematologic malignancies (including lymphoma, multiple myeloma)
* Prior RT of greater dose intensity than 100 Gy2 based on a biological effective dose (BED) calculation [BED (Gy2) = nd x (1+d/α/ß; where n=number of fractions, d=dose per fraction, α/ß=2)]
* Epidural tumor <2 mm from spinal cord
* Requirement of active receipt of systemic therapies concurrent with SBRT (concurrent hormonal therapies are allowed)
* Inability to lie flat and still for treatment delivery despite anti-anxiety and/or pain medications
* Non-English speakers are excluded from this study due to use of questionnaires which have not been validated in other languages.
* Patients lacking the capacity to describe their symptoms are excluded as that precludes them (or anyone on their behalf) from filling out the validated questionnaires about symptoms/toxicity.
* Pregnant women are excluded from this study because radiotherapy has the potential for teratogenic or abortifacient effects.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: if they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; or if diagnosed and treated within the past 2 years for cervical cancer in situ or basal cell or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2027-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Balboni, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oligometastatic Disease: Stereotactic Body Radiation Therapy (SBRT)to up to 3 sites of disease occurring in the bone or spine
  * Treatments will be delivered on a dedicated stereotactic linear accelerator that includes onboard conebeamCT imaging and orthogonal 2D/3D matching with robotic couch top.
  * Dosage will be determined by physician
  Stereotactic Body Radiation Therapy (SBRT)
  Stereotactic Linear Accelerator
- Re-irradiation to Metastatic Disease: Stereotactic Body Radiation Therapy (SBRT) to site(s) of disease occurring in the bone or spine
  * Treatments will be delivered on a dedicated stereotactic linear accelerator that includes onboard conebeamCT imaging and orthogonal 2D/3D matching with robotic couch top.
  * Dosage will be determined by physician
  Stereotactic Body Radiation Therapy (SBRT)
  Stereotactic Linear Accelerator
Period: Overall Study
Arm/Group | Oligometastatic Disease | Re-irradiation to Metastatic Disease
Started | 98 | 44 (The re-irradiation cohort is 44 instead of 50 because it excluded those who were lost to follow up and/or completed the surveys at time points different from protocol specified.)
Completed | 98 | 44 (The re-irradiation cohort is 44 instead of 50 because it excluded those who were lost to follow up and/or completed the surveys at time points different from protocol specified.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oligometastatic Disease | Re-irradiation to Metastatic Disease | Total
Number analyzed (Participants) | 98 | 44 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (10.4) | 61.5 (12.7) | 68.8 (NA) — SD was only calculated per cohort.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 10 | 90
  Male | 18 | 34 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 87 | 37 | 124
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: The 6-month Local Control Rate of SBRT
Description: The 6-month local control rate is the proportion of patients free of local failure at 6 months after stereotactic body radiation therapy (SBRT). Local failure is defined as the presence of biopsy-proven recurrence or radiologic scans that demonstrate progression at the treated sites.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Oligometastatic Disease | Re-irradiation to Metastatic Disease
Number analyzed (Participants) | 98 | 44
Participants | 94 | 40

2. Secondary Outcome: Number of Participants With 1-year Local Progression-Free Survival
Description: The local progression-free survival is defined as the duration of time from registration to time of local failure or death.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Oligometastatic Disease | Re-irradiation to Metastatic Disease
Number analyzed (Participants) | 98 | 44
Participants | 82 | 40

3. Secondary Outcome: Number of Participants With 2-year Progression-Free Survival
Description: Progression-free survival is defined as the duration of time from registration to time of any progression or death.
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Oligometastatic Disease | Re-irradiation to Metastatic Disease
Number analyzed (Participants) | 98 | 44
Participants | 46 | 16

4. Secondary Outcome: 2-year Overall Survival Rate
Description: Overall survival is defined as the time between registration and death.
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Oligometastatic Disease | Re-irradiation to Metastatic Disease
Number analyzed (Participants) | 98 | 44
Participants | 86 | 22

5. Secondary Outcome: Patient Reported Quality Of Life - Acute
Description: Patient reported QOL, symptoms and satisfaction will be assessed using the MDASI general questionnaire at baseline, during treatment and all follow-up visits.
Time Frame: 3 months
Reporting Status: Not Posted

6. Secondary Outcome: Patient Reported Quality of Life - Chronic
Description: as for outcome 5
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Post-baseline throughout protocol follow-ups. Maximum 5 years.
Description: CTEP Active Version of the NCI Common Terminology Criteria for Adverse Events (CTCAE)
Arm/Group | Oligometastatic Disease | Re-irradiation to Metastatic Disease
All-Cause Mortality (participants affected / at risk) | 28/98 | 29/44
Serious Adverse Events (participants affected / at risk) | 2/98 | 1/44
Other Adverse Events (participants affected / at risk) | 27/98 | 41/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oligometastatic Disease (N=98) | Re-irradiation to Metastatic Disease (N=44)
Atrial Fibrillation (Cardiac disorders) | 1 | 0 — Patient presented with new onset atrial fibrillation with a rapid ventricular response after receiving his chemotherapy regimen. He was treated with an IV of diltiazem, and prescribed heparin and coumadin after consult.
Hospitalization due to pain at an unrelated metastatic site (Musculoskeletal and connective tissue disorders) | 0 | 1 — Patient returned for protocol treatment and reported having increasing groin pain for 4 weeks. CT scan showed an increased left illiac bone lesion causing cortical destruction.
Prolonged hospitalization/Severe esophagitis (Gastrointestinal disorders) | 1 | 0 — Patient developed severe esophagitis requiring hospitalization and IV fluids over several days (grade 3). His symptoms improved with opioid medication optimization and he was discharged several days later.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oligometastatic Disease (N=98) | Re-irradiation to Metastatic Disease (N=44)
Fatigue (General disorders) | 10 | 24
Gastrointestinal (Gastrointestinal disorders) | 15 | 11
Pain (General disorders) | 7 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT02880319/Prot_SAP_000.pdf